CLINICAL TRIAL: NCT03499262
Title: Group Social ABCs: Early Intervention for Toddlers With Suspected ASD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Holland Bloorview Kids Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Jessica Brian, Clinical Psychologist, Holland Bloorview Kids Rehabilitation Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-745
Record Dates: First submitted 2018-02-22; First posted 2018-04-17 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Autism Spectrum Disorder; Autism
Keywords: Social ABCs; Early Intervention; Autism Spectrum Disorder (ASD); Toddler; Pivotal Response Treatment (PRT); Group Intervention; Parent-Mediated; Caregiver-Mediated; Social Communication; Positive Affect; Social Smiling; Social Orienting; Naturalistic Developmental Behaviour Intervention; NDBI; Autism; Early Identification
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Communication

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group Social ABcs (Experimental): Participants receiving Group Social ABCs intervention
  Interventions: Behavioral: Group Social ABCs

INTERVENTIONS:
Behavioral: Group Social ABCs — Social ABCs coach will facilitate the intervention to small groups of parents in a clinic setting, rather than the family's home. This new format allows the program to be completed in 6 weeks, versus the current 12-week model, and also offers the potential benefit of creating a parent support network within the program. Parents will still get live, one-on-one coaching for strategies to use with their child over the course of the program.

SUMMARY:
The Social ABCs is an evidence-based, developmentally informed, caregiver-mediated behavioural intervention for toddlers with suspected or confirmed Autism Spectrum Disorder (ASD). It is based on principles of Pivotal Response Treatment (PRT, grounded in Applied Behavioural Analysis), and responsive parenting. The two key targets of this program are functional verbal communication and positive caregiver-child affect sharing. This intervention takes place in the context of play and daily routines, and in all contexts is made to be fun.

In both a pilot study and a recently completed randomized control trial, toddlers whose caregivers received training in the Social ABCs intervention showed significant gains in early language development (both responsivity and initiations), increased child smiling (mediated by parent smiling), and a trend toward increased social orienting (one important manifestation of social attention).

In an effort to make the Social ABCs more feasible for community service providers to provide this intervention to higher number families, an abbreviated version of the Social ABCs intervention is being offered in a mixed group/individual format in a clinic setting. The primary goal of this pilot project is to assess feasibility of this abbreviated program in the novel format and setting. The secondary goal is to train clinical service providers to facilitate this intervention, thus introducing the program into community practice.

DETAILED DESCRIPTION:
The Social ABCs intervention was developed to meet the need for evidence-based, feasible, and sustainable interventions for toddlers with emerging ASD. Unlike other more comprehensive programs, the Social ABCs selectively targets only two key developmental areas (i.e., functional spoken language and positive affect). These domains were selected in order to promote developmental progress in areas thought to be central at this developmental stage in ASD. By targeting only two core domains, this program maximizes feasibility and portability (i.e., reduces resource demand) while effecting meaningful change with potential for collateral effects in untargeted, but related, areas.

Bolstered by evidence of acceptability, feasibility, and promise from a pilot study, the Social ABCs was subsequently evaluated in a large two-site RCT, demonstrating the efficacy of this caregiver-mediated intervention for toddlers with suspected or confirmed ASD. This study found child-level increases in vocal responsiveness, vocal initiations, child and parent smiling, and a trend toward increased social orienting in toddlers with suspected or confirmed ASD. Findings also demonstrated that caregivers attained fidelity relatively quickly, rated the intervention as highly acceptable, reported increased feelings of self-efficacy, and did not report increased stress associated with the burden of learning and providing the intervention.

Although the original Social ABCs model has demonstrated positive outcomes for children and their caregivers, it requires a large time commitment from both the Social ABCs coach and the family. Because of this, only a small number of children can receive the intervention at any given time in the original program. Given the urgent need for access to early interventions in ASD, a modified version of the Social ABCs ("Group Social ABCs") will be piloted and evaluated in order to increase access for more families in the community than the existing Social ABCs model. This new model has been carefully adapted to reach more families without sacrificing the meaningful aspects of the program.

In the Group Social ABCs project, the Social ABCs intervention itself remains the same as previous versions in terms of targeted skills, content, the parent coaching manual, and evaluation of fidelity and child responsivity. The difference is specifically in the delivery format. While the standard Social ABCs model was designed to be delivered exclusively in families' homes over a 12-week period, the Group Social ABCs model is shortened to 6 weeks and incorporates group informational sessions at Holland Bloorview along with some individualized live coaching sessions that also occur in clinic. By condensing the length of the program, incorporating group sessions, and offering this as a clinic-based program, the researchers hope to provide an intervention that is comparable in efficacy but able to reach a larger number of children than the original model.

Specifically, a Social ABCs coach will facilitate the intervention to small groups of 3-5 parents at a time in a clinic setting*, rather than the family's home. This new format allows the program to be completed in 6 weeks, versus the current 12-week model, and also offers the potential benefit of creating a parent support network within the program. Parents will still get live, one-on-one coaching for strategies to use with their child over the course of the program.

*In response to the 2020 global COVID-19 pandemic, study activities including both the group didactic and individual coaching sessions have shifted to an online format, with sessions being completed virtually. The protocol, delivery schedule, and session design remain the same. Baseline and follow-up data collection take place via mail and recorded video teleconference.

This project is highly relevant to early intervention, and thus outcomes, for children with ASD. This study has the potential to validate a model that will increase access to the Social ABCs for a greater number of families than the original program and will be more accessible to busy families who may not have had time for the original program. This means families who would otherwise not be able to access early intervention will now be able to participate.

The primary objective of this pilot study is to understand the impact of the Social ABCs in a condensed group format on child and caregiver outcomes, such as children's vocal communication, children's shared smiling with a caregiver, and caregiver implementation fidelity. The secondary objective is to identify any differences in the current project from previous Social ABCs findings. This may include child and/or caregiver outcomes as well as caregiver feelings of satisfaction with the Social ABCs training.

The primary hypothesis predicts that vocal responsivity to caregiver prompts will increase over the course of training. Secondary hypotheses predict the following will increase over the course of the training: child-initiated vocalizations, positive emotion sharing with a caregiver, orienting to caregiver, and caregiver fidelity of implementation.

ELIGIBILITY:
Inclusion Criteria:

* The child is a client of Holland Bloorview Kids Rehabilitation Hospital
* The child has clinically significant concerns of ASD
* The child participates in a maximum of 1 hour per week (monthly average) of the following interventions: speech/language, occupational, infant development, and physical therapy, and the family agrees to maintain this limit for the study duration
* The child's diet and medications are stable prior to starting the study, with plans to maintain relatively constant throughout the study.
* The caregiver is conversant in English and could be coached in English

Exclusion Criteria:

* The child has other neurological disorders or genetic syndromes that have known association with ASD (e.g., Fragile X syndrome)
* The child has significant uncorrected sensory impairments (vision, hearing, etc.)
* The child was born preterm (before 36 weeks' gestation)
* The child is experiencing an active regression of skills
* The child is involved in other behavioural interventions, such as ABA/IBI and the Hanen programs
* The child's diet and medications are undergoing drastic changes
* The caregiver has previously been trained in the Social ABCs or other PRT-based intervention program

Ages: 12 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 93 (Actual)
Dates: Start 2018-03-26 (Actual); Primary Completion 2020-12-23 (Actual); Study Completion 2020-12-23 (Actual)

PRIMARY OUTCOMES:
Vocal Responsivity | Baseline, Week 6
  Change in proportion of appropriate child vocal responses following a caregiver prompt in 10-minute video observation

SECONDARY OUTCOMES:
Vocal Initiations | Baseline, Week 6
  Change in rate of appropriate child-initiated vocalizations (Initiations); number per minute
Social Orienting | Baseline, Week 6
  Change in percentage of intervals with instances of social orienting (child looking at parent) per 10-minute video observation
Caregiver Fidelity of Implementation | Baseline, Week 6
  Change in percent of correct strategy implementation by parents (Fidelity) per 10-minute video observation

CONTACTS AND LOCATIONS:
Overall Officials: Jessica A Brian, PhD, Principal Investigator — Holland Bloorview Kids Rehabilitation Hospital
Locations (1):
- Holland Bloorview Kids Rehabilitation Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brian JA, Smith IM, Zwaigenbaum L, Bryson SE. Cross-site randomized control trial of the Social ABCs caregiver-mediated intervention for toddlers with autism spectrum disorder. Autism Res. 2017 Oct;10(10):1700-1711. doi: 10.1002/aur.1818. Epub 2017 Jun 2. PMID 28574669
- [Background] Brian JA, Smith IM, Zwaigenbaum L, Roberts W, Bryson SE. The Social ABCs caregiver-mediated intervention for toddlers with autism spectrum disorder: Feasibility, acceptability, and evidence of promise from a multisite study. Autism Res. 2016 Aug;9(8):899-912. doi: 10.1002/aur.1582. Epub 2015 Dec 21. PMID 26688077
- [Background] Landry SH, Smith KE, Swank PR. Responsive parenting: establishing early foundations for social, communication, and independent problem-solving skills. Dev Psychol. 2006 Jul;42(4):627-42. doi: 10.1037/0012-1649.42.4.627. PMID 16802896
- [Background] Brian JA, Bryson SE, Zwaigenbaum L. Autism spectrum disorder in infancy: developmental considerations in treatment targets. Curr Opin Neurol. 2015 Apr;28(2):117-23. doi: 10.1097/WCO.0000000000000182. PMID 25695137
- [Background] Zwaigenbaum L, Bryson S, Rogers T, Roberts W, Brian J, Szatmari P. Behavioral manifestations of autism in the first year of life. Int J Dev Neurosci. 2005 Apr-May;23(2-3):143-52. doi: 10.1016/j.ijdevneu.2004.05.001. PMID 15749241
- [Background] Smith IM, Koegel RL, Koegel LK, Openden DA, Fossum KL, Bryson SE. Effectiveness of a novel community-based early intervention model for children with autistic spectrum disorder. Am J Intellect Dev Disabil. 2010 Nov;115(6):504-23. doi: 10.1352/1944-7558-115.6.504. PMID 20946003